CLINICAL TRIAL: NCT02799407
Title: Electronic Consent of Numerous Subjects Employing Novel Techniques Trial
Acronym: ECONSENT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Never initiated.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00070430
Record Dates: First submitted 2016-06-06; First posted 2016-06-14 (Estimated); Last update posted 2024-04-12 (Actual); Status verified 2018-05

CONDITIONS: Informed Consent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Long Form Consent (No Intervention): Participants will receive the traditional long-form consent form.
- ResearchKit Consent (Experimental): Participants will receive the Apple ResearchKit consent form.
  Interventions: Other: ResearchKit Consent

INTERVENTIONS:
Other: ResearchKit Consent — Multi-tiered consent form using the Apple ResearchKit Platform.
  Arms: ResearchKit Consent

SUMMARY:
The purpose of this study is to compare the modular, multi-tiered consent process featured in Apple's ResearchKit (RK) to the standard consent process. The primary objective is to determine whether participants using the ResearchKit consent form have a significantly higher comprehension of the elements of consent than participants using the standard consent form.

DETAILED DESCRIPTION:
The purpose of this study is to compare the modular, multi-tiered consent process featured in Apple's ResearchKit (RK) to the standard consent process. The primary objective is to determine whether participants using the ResearchKit consent form have a significantly higher comprehension of the elements of consent than participants using the standard consent form. Through this two-arm randomized controlled trial (RCT) 120 participants will be asked to read through either a ResearchKit multi-tiered consent form administered on an iPod Touch device or a standard long-form consent form administered via paper and give their informed consent for a sham research study on health tracking apps. The participants will then be asked to answer a short series of questions (5 minutes) about the consent process in order to measure their subjective and objective comprehension. The main risk from this study is loss of confidentiality of responses, however this risk should be minimal given that protected health information (PHI) will only be collected on the consent document and all information will be stored on Duke Box in a private folder only accessible by the study team.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Able to read and understand study materials which are presented in English
* Owns or has access to a smartphone or other smart device such as a tablet or iPod

Exclusion Criteria:

* Any physical limitations which prevent the participant from using mobile and/or touch screen technologies
* Employed in a research position, clinical care position, or position which has regular exposure to clinical research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Participant comprehension, as measured by Qualtrics survey | at study conclusion, an average of 15 minutes
  Participants will complete a questionnaire about the consent form after reading through the consent which will assess their comprehension of the contents of the consent process.

CONTACTS AND LOCATIONS:
Overall Officials: David Tanaka, MD, Principal Investigator — Duke Health

IPD SHARING:
Plan to Share IPD: No